CLINICAL TRIAL: NCT00012948
Title: Centralized Telephone Outreach to Assist Smoking Cessation Among Veterans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: SUI 99-101
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Telephone Care

INTERVENTIONS:
Procedure: Telephone Care

SUMMARY:
Smoking cessation interventions including behavioral and pharmacological components have been demonstrated to be both effective and cost-effective. Although there is a high prevalence of smoking and smoking-related disorders among veterans who use VA medical centers for health care, rates of identification of tobacco use and provision of brief and/or intensive smoking cessation services are suboptimal. Telephone outreach (TO) may serve to increase access to counseling and medications to assist smoking cessation. From the standpoint of health systems, TO provides the opportunity for centralized oversight and quality assurance, economy of scale, and dissemination strategies that are practical to implement. At the provider level, TO addresses barriers to delivery of services such as limited time and skills. From the standpoint of the smoker, attractions of TO include accessibility, convenience, and privacy.

DETAILED DESCRIPTION:
Background:

Smoking cessation interventions including behavioral and pharmacological components have been demonstrated to be both effective and cost-effective. Although there is a high prevalence of smoking and smoking-related disorders among veterans who use VA medical centers for health care, rates of identification of tobacco use and provision of brief and/or intensive smoking cessation services are suboptimal. Telephone outreach (TO) may serve to increase access to counseling and medications to assist smoking cessation. From the standpoint of health systems, TO provides the opportunity for centralized oversight and quality assurance, economy of scale, and dissemination strategies that are practical to implement. At the provider level, TO addresses barriers to delivery of services such as limited time and skills. From the standpoint of the smoker, attractions of TO include accessibility, convenience, and privacy.

Objectives:

The objectives of the study are to: 1) determine if TO increases successful quitting among veterans who smoke, compared to the distribution of written self-help materials; and 2) determine the cost-effectiveness of TO for smoking cessation for veterans who smoke.

Methods:

The study involved a population-based sample of veterans in VISN 13 who use one of the five Network VAMCs for primary care. 838 smokers were recruited, enrolled and randomly assigned to 1) written self-help materials + TO, or 2) written self-help materials alone. The behavioral intervention protocol included follow-up calls scheduled in a relapse-sensitive fashion. Use of nicotine replacement therapy (NRT) was encouraged, and prescriptions facilitated. Data was collected at baseline, 3 months, and 12 months by telephone. Information on demographic characteristics, medical and mental health histories, smoking history, intervention, and use of clinical services for smoking cessation was included. Cost data will be calculated from administrative databases, and will include 1) written materials, 2) counseling (personnel time, equipment, space), and 3) medications. The primary outcome was 6 months of prolonged abstinence from smoking, measured 12 months following intervention. Secondary analyses evaluated 3 month and 12 month point prevalent abstinence from smoking, quit attempts, and a formal cost-effectiveness analysis that will include total costs, total and marginal effects and cost-effectiveness ratios (average cost/quit and average cost/marginal quit) for TO and SH interventions.

Status:

Data collection and main outcome analyses have been completed. The main manuscript will be submitted to JAMA in October 2004. We are starting cost-effectiveness analyses.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be smokers who have a phone and who speak English. They are excluded for psychiatric instability.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne M. Joseph, MD MPH, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] An LC, Zhu SH, Nelson DB, Arikian NJ, Nugent S, Partin MR, Joseph AM. Benefits of telephone care over primary care for smoking cessation: a randomized trial. Arch Intern Med. 2006 Mar 13;166(5):536-42. doi: 10.1001/archinte.166.5.536. PMID 16534040